CLINICAL TRIAL: NCT01316198
Title: Alteration of Optical Density and Plasma Xanthophylls After Short Term Supplementation With Macular Carotenoids in Patients With AMD
Brief Title: Effects of Xanthophylls on Optical Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Volker Boehm, Dr. Volker Böhm, University of Jena
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BioPlant-LZ-AMD2011
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Age-Related Macular Degeneration
Keywords: human study; AMD; lutein; zeaxanthin; optical density
MeSH Terms: conditions — Macular Degeneration | interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lutein and zeaxanthin (Experimental)
  Interventions: Dietary Supplement: Verum
- Placebo (Experimental)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Verum — 10 subjects consume for 4 weeks a beverage containing 10 mg lutein and 3 mg zeaxanthin per day
  Arms: Lutein and zeaxanthin
Dietary Supplement: Placebo — 10 subjects consume for 4 weeks a placebo beverage without any lutein and zeaxanthin
  Arms: Placebo

SUMMARY:
The objective of the study was to investigate the influence of a intervention with lutein und zeaxanthin from crucifers on the optical density of the macular pigment of patients with non exudative age-related maculopathy. It is hypothesized that the applied study beverage elevates plasma concentrations of the administered xanthophylls and the optical density after 4 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients with non exudative age-related maculopathy

Exclusion Criteria:

* intake of dietary supplements containing lutein and zeaxanthin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Optical density of macular pigment in AMD patients | 10 weeks

SECONDARY OUTCOMES:
Concentration of xanthophylls in plasma of AMD patients | 10 weeks
blood lipids | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Volker Boehm, Dr., Principal Investigator — Friedrich Schiller University Jena, Institute of Nutrition, RG Bioactice Plant Products
Locations (1):
- Friedrich Schiller University, Jena, Thuringia, Germany